CLINICAL TRIAL: NCT04109430
Title: Study of PtiO2 Variation by Body Temperature and Capnia in Severe Head Trauma Patients With Intracranial Refractory Hypertension Treated With Targeted Temperature Control
Brief Title: Study of PbiO2 Variation by Body Temperature and Capnia in Severe Head Trauma Patients Treated With Targeted Temperature Control
Acronym: TODAY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TODAY STUDY (29BRC19.0064)
Record Dates: First submitted 2019-09-19; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Severe Brain Injury
Keywords: PbtO2; hypothermia; trauma brain injury; targeted control temperature; refractory brain hypertension
MeSH Terms: conditions — Brain Injuries; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Serious head trauma is a common and pathology and responsible of high morbidity and mortality. The major challenge, from the very first hours, is to limit cerebral ischemia by controlling secondary brain injury factors.

These parameters must be integrated early in order to guide the better cerebral resuscitation. Brain monitoring is multimodal:transcranial Doppler, intracranial pressure sensor, cerebral tissue pressure in O2.

In the case of refractory intracranial hypertension to well-conducted medical treatment, targeted temperature control showed its efficacy on the control of intracranial pressure.

There are few data in the literature on PbtO2 modifications during therapeutic hypothermia.

PbtO2 monitoring is now commonly used according to literature data, showing the benefit of the latter but the interpretation of its values during the phase of targeted temperature control is not known. Due to the lack of data on the variation of values of PbtO2 during the hypothermia phase, values falsely comfortable or falsely weak could lead respectively to a lack of support of an episode of tissue hypoxia or the introduction of unjustified aggressive therapeutics.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, mono-centric study at surgical intensive care unit at Brest medical university hospital.

This study will be conducted in a reference center for the management of patients with traumatic brain injury, who is used to collect prospective data.

The clinical research structure of Brest Medical University allows data analysis and the investigators have the clinical knowledge for their interpretation.

After verification of the inclusion and non-inclusion criteria and information of the family (parent or relative) or the holder of parental authority, patients will be included in order of arrival in the service.

The population studied is the trauma brain injured patients with an initial Glasgow coma scale of less than 8 at pre-hospital care or neurological impairment with Glasgow Coma Scaleless than 8 in the first 24 hours after admission to intensive care.

The installation of a intra-cranial pressure/ PbtO2 probe (INTEGRA Licox PtO2 monitor) is performed by the neurosurgeon according to the protocol service.

Approximately 30 patients were monitored with a PbtO2 sensor in 2018 in the Surgical intensive care unit at Brest Medical University Hospital.

After verification of inclusion and non-inclusion criteria, oral and written information will be given to parent or relative of the patient. A no-objection form will be sent to the patient as soon as possible to confirm his participation.

Follow-up of the patient is carried out until discharge of intensiv care unit. The duration of participation in the study is the duration of treatment by targeted temperature control, very variable depending on the clinical evolution of patients, from 1 day to more than one week. The management of the patients included in this study is not modified in relation to the treatment usually recommended in the intensiv care unit.(based on French recommendation).

In order to describe the variations of PbtO2 values, the PbtO2 values are collected at time T0 before induction of targeted temperature control, at time T1: the first hour of the targeted temperature control phase (<35 ° C) at time T2: during the phase of temperature stability (<35 ° C) defined as two successive hours of hypothermia, at time T3 defines as 6 hours at a stable temperature in hypothermia, then once a day up to the end of the targeted temperature control phase.

Then the values of PtiO2 are collected during the daily hypercapnia test during targeted temperature control phase.

Demographic data collected are age, sex, weight, height, and data on gravity at the entrance: IGS2 score, first Glasgow Coma scale score, time to CT-scan and IMPACT score.

Data on time to PbtO2 probe and ICP probe insertion and time to equilibration of PbtO2 value.

Data were collected at all times, T0, T1, T2, T3 (as defined above) and daily: the body temperature (collected by esophageal thermal probe), the cerebral perfusion pressure, the value of PtiO2 / PIC, FiO2 / etCO2, an arterial blood sample, a blood count and a daily ionogram,daily transcranial Doppler data, doses of amines, curares and sedation.

During the stay were collected: time to and nature of the surgical procedure and realization of a craniectomy or not, position of the PtiO2 probe on a control scanner, an at the discharge: prognosis score (GOS-E),lenght of stay in intensive care unit, death in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* age> 15 years
* severe traumatic brain injury defined by an initial Glasgow Coma Scale score less than 8 or neurological impairment in the first 24 hours with Glasgow less than 8,
* brain hypertension refractory despite usual sedation and control of ACSOS (ICP> 20mmHg for more than 15 minutes over a period of one hour)
* Participation Agreement.

Exclusion Criteria:

* initial bilateral mydriasis
* no information of the family
* refusal of participation.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Organized and practiced on the human being for the development of biological and medical knowledge, in which the acts are practiced and the products used in the usual way, without additional or unusual procedure of diagnosis, treatment or monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in PbtO2 gross values during the targeted temperature control phase | 1 year (through study completion)
  Evaluated at the time T0 before induction of the targeted control of the temperature, at time T1: the first hour of the targeted temperature control phase (<35 ° C), at time T2: during the stability phase of the temperature (<35 ° C) defines as two successive hours of hypothermia, at time T3 defines as 6 hours at a stable temperature under hypothermia, then once a day until the control phase targeted temperature stops.

SECONDARY OUTCOMES:
Changes in PtiO2 gross values during hypercapnia test | 1 year (through study completion)
  Description of variations values of PbtO2 during hypercapnia test induced by ventilation minute reduction, performed to assess brain tolerance to possible warming.

CONTACTS AND LOCATIONS:
Locations (1):
- HUET, Brest, Brittany Region, France